CLINICAL TRIAL: NCT07168408
Title: Procedural Skills Transfer in Bronchoscopy
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: R&D 2021/0163
Record Dates: First submitted 2024-07-17; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Up to 300 patients undergoing routine bronchoscopy procedures. Patients will be asked permission to access previous CT scans and record video from the bronchoscopy procedure.
- Group 2: Up to 20 bronchoscopists. These participants will be asked a to complete a short questionnaire on their experience and will wear a sensorized glove to capture their hand movements during the procedure

SUMMARY:
Brief summary The goal of this Feasibility study is to capture bronchoscopy data from patients (Group1) and bronchoscopists (Group 2) over a period of three years. The investigators wish to collect the pre-procedure CT scans and endoscopy videos of 300 patients. Up to 20 bronchoscopists will take part in the study

Primary outcomes

1. To collect imaging data from patients undergoing routine bronchoscopy procedures
2. To collect movement data from clinicians performing the routine bronchoscopy procedures using a sensory Glove

Secondary outcomes

1. Integrate the data gathered with procedure guidelines to develop a representation of procedure success using machine learning algorithms.
2. Develop an actionable knowledge base for bronchoscopy skill transfer to novice/untrained medical staff.
3. Investigate the feasibility of developing models of bronchoscopy procedures to develop training tools in the future

There are no additional samples or time commitments from the participants in Group 1.

The participants in Group 2 will be asked to answer a short questionnaire about their experience in performing bronchoscopies and will be asked to wear a sensory glove during the bronchoscopy procedure to capture their hand movements.

DETAILED DESCRIPTION:
Bronchoscopy is a procedure for visualising the inside of the lung and airways. During bronchoscopy, a thin tube is passed through the patient's mouth or nose, down the throat and into the lungs. This allows the practitioner to examine the patient's airways for abnormalities such as inflammation. Additionally, samples may be taken from inside the lungs.

Success rate of bronchoscopy relies on the practitioners experience. Patients undergoing bronchoscopy performed by novice bronchoscopists have an increased complication rate. Data from clinical practice suggest that bronchoscopy has a prolonged learning curve and trainees should perform a number of procedures, under supervision, to learn the technique.

In this study the investigators aim to capture bronchoscopy data from patients (Group1) and bronchoscopists (Group 2) over a period of 3 years. The investigators will collect the pre-procedure CT scans and endoscopy videos of 300 patients. Up to 20 bronchoscopists will take part in the study by answering a short questionnaire on their experience and wearing sensorized gloves which will record their hand movements during the procedure. the investigators aim to use this data to develop computer algorithms and simulators that will assist in the training of new bronchoscopists, decreasing the time required to learn the technique and improving patient safety.

ELIGIBILITY:
Inclusion Criteria Group 1

* over 16 years of age
* patients identified as requiring a bronchoscopy by their clinician
* patients must have had a CT scan in the 8 weeks prior to the procedure
* capacity to consent

Exclusion Criteria Group 1 - Patients who have not had a CT scan in the 8 weeks prior to the procedure

Inclusion Criteria Group 2

- Suitably qualified bronchoscopists, this may include trainee bronchoscopists

Exclusion Criteria Group 2

* Clinicians who do not give consent to participate in the study
* Clinicians who are not comfortable performing bronchoscopy while wearing the lightweight glove

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group 1- Patients undergoing a routine, clinically indicated bronchoscopy procedure
  Group 2- Clinicians currently involved in performing bronchoscopy procedures
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To collect imaging data from patients undergoing routine bronchoscopy procedures | up to 1 hour
  The bronchoscopy images will be recorded using a screen capture device
to collect movement data from clinicians performing the routine bronchoscopy procedures | up to 1 hour
  A sensory glove will be worn by the clinicians to capture their hand movements during the routine bronchoscopy

SECONDARY OUTCOMES:
Integrate the data gathered with procedure guidelines to develop a representation of procedure success using machine learning algorithms | 1 year after completion of data collection
  Develop machine learning algorithms to
Investigate the feasibility of developing models of bronchoscopy procedures to develop training tools in the future. | 1 year after completion of data collection
  Once data has been analysed investigate whether this can be used to develop training tools for future clinicians

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data generated by the study (including personal data) will not be transferred to external individuals or organisations outside of the sponsoring organisations